CLINICAL TRIAL: NCT05008965
Title: A Phase II Study to Evaluate the Efficacy and Safety of FB825 in Adult Patients With Moderate-to-severe Allergic Asthma
Brief Title: Evaluate the Efficacy and Safety of FB825 in Adult With Allergic Asthma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Oneness Biotech Co., Ltd. (Industry)
Collaborators: Microbio Shanghai Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FB825CLCT03
Record Dates: First submitted 2021-02-13; First posted 2021-08-17 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Allergic Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FB825 (Experimental)
  Interventions: Drug: FB825
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FB825 — FB825 will be administered at 8 mg/kg for the first dose and 4 mg/kg for the other five doses.
  Arms: FB825
Drug: Placebo — Placebo will be administered at 8 mg/kg for the first dose and 4 mg/kg for the other five doses.
  Arms: Placebo

SUMMARY:
This is a randomized, placebo-controlled and double-blind study to evaluate the efficacy and safety of FB825 in adult patients with moderate-to-severe allergic asthma.

DETAILED DESCRIPTION:
The study comprises of a 4-week screening period, a 24-week treatment period and a 12-week follow-up period.

It is anticipated that approximately 100 subjects will be enrolled into this trial, in order to complete a total of 92 evaluable subjects. Eligible subjects will be randomized to receive placebo or FB825 in a 1:1 ratio.

Eligibility will be checked in patients with allergic asthma during the 4-week screening period. Potential candidates should provide signed informed consent forms before starting any screening activities. The subjects will receive one dose of 8 mg/kg FB825 or placebo, and five doses of 4 mg/kg FB825 or placebo every 4 weeks subsequently. The study drug will be administered as a 1-hour IV infusion.

Patients may administer albuterol (or equivalents) as rescue medications as needed throughout the study.

Prior to screening, patients must be on a stable dose of any of formulations of ICS/LABA combination therapy for at least 1 month. Patients who have been on medium to high dose medication according to the GINA guidelines (GINA, 2021) maintained at randomization (Day 1) will remain on their current treatment as background therapy.

ICS/LABA combination therapy during background therapy stable phase (Day -28 to Day 28) followed by ICS (fluticasone or equivalent) during ICS tapering phase (Day 29 to Day 112 or Day 140), and then followed by the FB825 monotherapy phase (Day 113 or Day 141 to Day 168).

Upon completing 24 weeks of treatment with the investigational product, patients will be placed on ICS/LABA combination therapy and albuterol (or equivalents) (as needed) to control their symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Male or females 18-75 years old.
2. Subjects diagnosed with moderate-to-severe allergic asthma [Global Initiative for Asthma [GINA]; GINA, 2021) at least 12 months prior to Visit 1.
3. Documented reversibility from historical data of at least 12% and 200 mL in FEV1 after the administration of 200 to 400 mcg albuterol/salbutamol (or other standard office practice) OR documented airway hyperresponsiveness (methacholine PC20 < 8 mg/mL [or PC20 < 16 mg/mL on ICS]) OR airflow variability in clinic FEV1 >12% and 200 mL between visits outside of respiratory infections, documented in the past 24 months prior to Visit 1 if documented reversibility and airway hyperresponsiveness data are not available.
4. Subjects must have a pre-bronchodilator FEV1 value of ≥ 40% and ≤ 80% predicted within 2 months from randomization.
5. Subjects must have received a physician-prescribed asthma regimen with medium- or high-dose ICS plus LABA for at least 3 month prior to Visit 1 and the dose of ICS must be stable for at least 30 days prior to Visit 1 and throughout the screening period.

   1. High-dose ICS is defined as total daily dose of >500 mcg fluticasone propionate or equivalent
   2. Medium-dose ICS is defined as a total daily dose of 250 to 500 mcg fluticasone propionate or equivalent.
   3. Equivalence ICS doses will be based upon the GINA guidelines (GINA, 2021)
   4. According to the medical history, subject have no more than a maximum of 2000 mcg/day equipotent ICS daily dosage of fluticasone propionate or equivalent in 3 months before visit 1.
6. Prior to screening, subjects must be on a stable dose of any of the following doses and formulations of ICS/LABA combination therapy for at least 1 month:

   1. Fluticasone/salmeterol combination therapy

      * Advair® Diskus - dry powder inhaler (DPI): 250/50 μg BID or 500/50 μg BID, or
      * Advair® HFA - metered dose inhaler (MDI): 230/42 μg BID or 460/42 μg BID, or
   2. Budesonide/formoterol combination therapy (Symbicort® -160/4.5 μg BID or 320/9 μg BID), or
   3. Mometasone/formoterol combination therapy (Dulera® -200/10 μg BID or 400/10 μg BID).
   4. Other equivalents medium to-high dose medication following the GINA guidelines (GINA, 2021)
7. Subjects must have a documented history of protocol-defined asthma exacerbation at least 1 or more times within the 12 months.
8. A total serum IgE ≥ 125 IU/mL during screening prior to randomization.
9. Subjects must have at least one positive in skin prick test or at least one environmental allergen-specific IgE greater than normal range.
10. Uncontrolled asthma demonstrated both during the screening period and at the time of randomization defined as ACQ-5 (5-item Asthma Control Questionnaire) ≥ 1.5
11. If recently treated for respiratory tract infection, the treatment must have been completed at least 4 weeks prior to screening. Subjects who have an upper respiratory tract infection during screening are allowed to be rescreened 4 weeks after resolution.
12. Female subjects of childbearing potential must use at least two forms of birth control. One must be barrier protection (i.e., condom or female condom) and the other is one of acceptable method of birth control (ie, diaphragm, intrauterine device, hormonal contraceptives, or abstinence) throughout the study. Subjects who are surgically sterile (ie, hysterectomy, bilateral tubal ligation, or bilateral oophorectomy), or postmenopausal (defined as amenorrhea for 12 consecutive months and documented serum follicle stimulating hormone level >40 mU/mL) will be considered as no childbearing potential. All female subjects of child-bearing potential must have a negative serum pregnancy test at screening.

    Note: The subject must use the methods of contraception mentioned above during study period and at least 120 days after the last dosing of FB825.
13. The subject has a body weight ≥ 40 kg at screening.
14. The subject has a normal or non clinically significant abnormal, as determined by the investigator, 12-lead electrocardiogram (ECG).
15. The subject is able to provide written informed consent.
16. The subject agrees to comply with all protocol requirements.

Exclusion Criteria:

1. Asthma exacerbation or any other reason requiring systemic steroids in the 30 days prior to randomization. Subjects are allowed to be rescreened 30 days after completion of treatment.
2. >20% relative change in post-bronchodilator FEV1 between screening and randomization.
3. Female subjects who are pregnant or lactating.
4. A positive human immunodeficiency virus (HIV) test (e.g., HIV Ag/Ab combo test) at screening or subject taking antiretroviral medications, as determined by medical history.
5. Patients with positive HBeAg or HCV RNA results should be excluded as they are indications of active Hepatitis B virus and Hepatitis C virus replication.
6. Active lung diseases (e.g., bronchitis, chronic obstructive pulmonary disease) other than allergic asthma.
7. Use of any experimental drug within 30 days or 5 half-lives, whichever is longer, prior to or during the screening period.
8. Current or history of treatment with a monoclonal antibody, for example, IL-4, IL-5, IL-13 or IL-15 antibody treatment within 6 months prior to the screening.
9. Current or history of treatment with anti-IgE antibody treatment within 6 months or 5 half-lives, whichever is longer.
10. The subject has a history of alcohol or drug abuse that would impair or risk the patients' full participation in the study, in the opinion of the investigator.
11. The subject has any condition that, in the opinion of the investigator, would compromise the study or the well-being of the subject or prevent the subject from meeting or performing study requirements.
12. The subject has indication of severe liver disease, defined by serum levels of either alanine aminotransferase (ALT), aspartate transaminase (AST) above 3x upper limits of normal (ULN) or elevated total bilirubin >2x ULN as determined at screening.
13. The subject has severe kidney disease, defined as estimated GFR <30ml/min/1.73m2 or creatinine > 3x ULN.
14. The subject has known or suspected history of immunosuppression or immunodeficiency.
15. Known history of active tuberculosis (TB) or evidence of tuberculosis infection as defined by a positive purified protein derivative (PPD) skin test and/or interferon-gamma release assay. The interferon-gamma release assay should be repeated in case of an indeterminate result.
16. The subject has history of malignancy within 5 years before the screening period. Patients with non-invasive carcinoma in-situ of the cervix, basal cell carcinoma or squamous cell carcinoma of the skin may be eligible if they have undergone curative resection at least 12 months prior to screening.
17. Current smoker with > 10 packs year prior to screening. A smoker is defined as a subject who has taken inhaled nicotine containing products (e.g. cigarette, cigar, pipe), including e-cigarettes prior to screening.
18. High risk of parasite infection

    • Risk factors for parasitic disease (living in an endemic area, travel within the last 6 months to regions where geohelminthic infections are endemic, and/or chronic immunosuppression).

    AND

    • Evidence of parasitic colonization or infection on stool evaluation for ova and parasites.

    Note: stool ova and parasite evaluation will only be conducted in patients with risk factors and an eosinophil count more than twice the upper limit of normal.
19. The subject has received live vaccine within 12 weeks or COVID-19 vaccination within 2 weeks prior to dosing or planned live attenuated vaccinations during the study.
20. The subject has a history of any clinically relevant arrhythmias as determined by the investigator.
21. The subject has a history of respiratory failure or near fatal asthma events which resulted in intensive care unit admission or intubation within five years before the screening period.
22. History of anaphylaxis to any biologic therapy.
23. The subject has major surgery, for example organ replacement, joint replacement, full hysterectomy, heart surgeries, within 8 weeks before the screening. The subject who has major surgery prior to 8 weeks of screening should have fully recovered from any surgical procedures.
24. The subject has comorbid disease that might interfere with the evaluation of IMP (investigational medicinal product) or conduct of study procedures (eg, bronchodilator test).
25. The subject requiring non-selective beta-adrenergic receptor blockers for any reason and initiation or dose change of a selective beta-1 adrenergic receptor blocker within 3 months prior to Visit 1.
26. The subject who received bronchial thermoplasty within 3 years of Visit 1 OR patients who plan to begin therapy during the Screening Period or the Randomized Treatment Period.
27. The subject with active autoimmune disease (excluding atopic dermatitis) or patients using immunosuppressive therapy for autoimmune disease (excluding atopic dermatitis) (eg, rheumatoid arthritis, inflammatory bowel disease, primary biliary cirrhosis, systemic lupus erythematosus, multiple sclerosis, etc.) or patients with high titer autoantibodies at screening who are suspected of having high risk for developing autoimmune disease at the discretion of the Investigator or the Sponsor.
28. Use of Traditional Chinese Medications, those that are listed in the Prohibited Medication, for the treatment of asthma within 3 months prior to screening.
29. Aggravating factors that are inadequately controlled e.g., medication uncontrolled gastroesophageal reflux disease.
30. The subject has adrenal insufficiency (ACTH-resistant) by rapid ACTH stimulation test due to known history of adrenal insufficiency or being suspected of adrenal insufficiency or long-term use of systemic corticosteroids (annual average more than 6 months in the past two years).

    Adrenal insufficiency: after 30 minutes of ACTH injection, the cortisol level ≦20 mg/ml in rapid ACTH stimulation test.
31. History of prior positive SARS-CoV-2 diagnostic test (antigen or NAAT/PCR) within 3 months prior to screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-07-27 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of an exacerbation of asthma at week 24 after first dosing. | week 24

SECONDARY OUTCOMES:
Mean change in morning peak expiratory flow (PEF) from baseline | week 12, 16, and 24
Change in ACQ 5 from baseline | week 12, 16, and 24
Percentage of patients achieving decrease in score by greater than or equal to 0.5 points on the ACQ (with a minimal importance difference improvement) | week 12, 16, and 24
Change in FEV1 from baseline | week 12, 16, and 24
Occurrence of an exacerbation of asthma | week 12 and 16
The incidence of treatment emergent adverse events throughout the study | Week 24

OTHER OUTCOMES:
Change in Total IgE from baseline | week 12, 16, and 24

CONTACTS AND LOCATIONS:
Overall Officials: Sam Kuo, Principal Investigator — Oneness Biotech Co., Ltd.
Locations (13):
- Taiwan (13):
  - Kaohsiung Chang Gung Medical Foundation, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Far Eastern Memorial Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - Taichung Venterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Linkou Chang Gung Memorial Hospital, Taipei
  - MacKay Memorial Hospital, Taipei
  - Ministry of Health and Welfare Shuang-Ho Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Municipal Wanfang Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei